CLINICAL TRIAL: NCT02653729
Title: Cognitive Behaviour Therapy for Psychosis in First Episode Patient and the Outcome of Cognitive Behaviour Therapy on Psychotic Symptoms
Brief Title: Cbt for Psychosis and Affect on Psychosis Symptoms
Acronym: cbtpaps
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aisha Andleeb (Other)
Responsible Party: Sponsor-Investigator, Aisha Andleeb, M.phil Scholars Department of Applied Psychology, Bahauddin Zakariya University
Organization: Bahauddin Zakariya University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: abdulsattar
Record Dates: First submitted 2016-01-07; First posted 2016-01-12 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Psychosis
Keywords: cognitive behaviour therapy; first episode
MeSH Terms: conditions — Psychotic Disorders | interventions — Cognitive Behavioral Therapy; Psychotherapy; Rieske iron-sulfur protein; 24,25-oxidolanosterol; 2-((((2-chloroethyl)-nitrosoamino)carbonyl)amino)-1,3-cyclohexanediol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Espidone, Olepra, Donu & C.B.T (Experimental): Espidone tablet 2 mg and Donu 10 mg by mouth twice a day and Olepra tablet 5 mg by mouth at night and C.B.T 6 session program 45 minutes session after every 15 days
  Interventions: Behavioral: cognitive behaviour therapy; Drug: Espidone; Drug: Olepra; Drug: Donu
- Espidone, Olepra & Donu (Active Comparator): Espidone tablet 2 mg and Donu 10 mg by mouth twice a day Olepra tablet 5 mg by mouth at night
  Interventions: Drug: Espidone; Drug: Olepra; Drug: Donu

INTERVENTIONS:
Behavioral: cognitive behaviour therapy
  Other Names: talk therapy; conversation therapy
  Arms: Espidone, Olepra, Donu & C.B.T
Drug: Espidone
  Other Names: risp
Drug: Olepra
  Other Names: olan
Drug: Donu
  Other Names: zanzia

SUMMARY:
This study aims to examine the effectiveness of cognitive behavior therapy for psychosis in first episode patients and see the outcome of CBT on psychotic symptoms. Because cognitive behavior therapy mostly use in depressive patient to treat the negative thinking pattern Cognitive behavioral approaches in the treatment of psychosis have become more prevalent in recent years for a number of reasons. Evidence has been available for the past two or three decades regarding the success of these techniques with other forms of psychopathology such as depression, anxiety disorders, and medical problems. Anxiety, depression and low self-esteem have been cited as the most common consequences of psychotic disorders. The observation has also emerged that many patients develop their own coping strategies for reducing the frequency, severity, and disruptiveness of their symptoms. There has also been increasing evidence regarding the influence of social environmental factors on the course of psychosis and the development of stress-vulnerability models to explain these relationships. Research suggests that 20 to 50 percent of persons with psychosis who receive neuroleptics continue to experience difficulties related to their psychotic symptoms.

DETAILED DESCRIPTION:
This research aims to examine the effect of cognitive and behavior therapy for psychosis in first episode patients and see the outcome of CBT on psychotic symptoms.

Cognitive and Behavior Therapy for Psychosis

Cognitive behavioral therapy (CBT) is talking therapy that can help to manage problems by changing the way you think and behave.

There are notable clinical successes in treating common emotional disorders using cognitive-behavioral approaches based on precise theoretical models. In anxiety disorders, the underlying fear beliefs are tested in behavioral experiments to substantially reduce symptoms; in depression, mood is lifted by reevaluating negative views of the self and limiting excessive rumination.

With psychosis, similar psychological processes are active in the experience of delusions and hallucinations. For example, persecutory delusions are conceptualized as threat beliefs that are the patient's attempts to make sense of his or her personal experiences, while hallucinations are problematic when they are interpreted by the patient as representing powerful and destructive forces. Hence, in cognitive therapy for psychosis, fearful thoughts are carefully reevaluated; withdrawal from social contact and activity is gradually reversed; and feelings of hope, control, and self-worth are fostered. Patients with psychosis are given time to talk about their experiences and, importantly, strategies are developed from this collaborative discussion.

In this one-on-one therapy, distressing experiences take center stage. The first generation of cognitive-behavioral therapy (CBT) for psychosis, when added to standard care, has demonstrated efficacy in treating patients with delusions and hallucinations.

Psychosis Psychosis is a serious mental disorder characterized by thinking and emotions that are so impaired, that they indicate that the person experiencing them has lost contact with reality.

People with psychosis are described as psychotic. People experiencing psychosis may exhibit some personality changes and thought disorder. Depending on its severity, this may be accompanied by unusual or bizarre behavior, as well as difficulty with social interaction and impairment in carrying out daily life activities.

The term "psychosis" is very broad and can mean anything from relatively normal aberrant experiences through to the complex and catatonic expressions of schizophrenia and bipolar type 1 disorder. In properly diagnosed psychiatric disorders (where other causes have been excluded by extensive medical and biological laboratory tests), psychosis is a descriptive term for the hallucinations, delusions, sometimes violence, and impaired insight that may occur. Psychosis is generally the term given to noticeable deficits in normal behavior (negative signs) and more commonly to diverse types of hallucinations or delusional beliefs, especially as regards the relation between self and others as in grandiosity and paranoia.

Objectives

1. To explore the effect of cognitive behavior therapy for psychosis in first episode patients.
2. To develop a guide to conduct cognitive behavior therapy in early psychosis patients.
3. To evaluate the major clinical outcomes in the treatment of psychotic symptoms.
4. To examine the feasibility of cognitive behavior therapy in psychotic patients. Rationale of the study This study aims to examine the effectiveness of cognitive behavior therapy for psychosis in first episode patients and see the outcome of CBT on psychotic symptoms. Because cognitive behavior therapy mostly use in depressive patient to treat the negative thinking pattern

Cognitive behavioral approaches in the treatment of psychosis have become more prevalent in recent years for a number of reasons. Evidence has been available for the past two or three decades regarding the success of these techniques with other forms of psychopathology such as depression, anxiety disorders, and medical problems. Anxiety, depression and low self-esteem have been cited as the most common consequences of psychotic disorders. The observation has also emerged that many patients develop their own coping strategies for reducing the frequency, severity, and disruptiveness of their symptoms. There has also been increasing evidence regarding the influence of social environmental factors on the course of psychosis and the development of stress-vulnerability models to explain these relationships. Research suggests that 20 to 50 percent of persons with psychosis who receive neuroleptics continue to experience difficulties related to their psychotic symptoms.

The therapeutic process consists of helping the patient become aware of his or her internal stream of thoughts when distressed, and to identify and modify the dysfunctional thoughts. Behavioral techniques are used to bring about functional changes in behavior, regulate emotion, and help the cognitive restructuring process. Modifying the patient's underlying dysfunctional beliefs leads to lasting improvements. In this structured therapy, the therapist and patient work collaboratively to use an approach that features reality testing and experimentation.

Method

Research Design The present study will be a feasibility rater blind randomized controlled trial study to test the efficacy of brief CBT for patients with suffering from first episode psychosis.

Sample Total 50 patients meeting the inclusion criteria of the study will be recruited from psychiatry unit of a public hospital of Raheem yar khan, Pakistan. conducted by using 50 patient met the eligibility criteria.

Instruments/Assessment Measures

The following assessment measures will be used in the research:

1. The Psychotic Symptom Rating Scales.
2. Positive and Negative Symptom Scale.
3. Schedule for Assessment of Insight.

Procedure

1. Authors of scales will be informed about usage of the scale in current research.
2. Get permission to Dr.Farooq Naeem usage of the CBT manual of psychosis.
3. SPSSv.20 for data analysis

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with psychosis by psychiatrist of the recruiting unit.
* Patients with duration of illness till 3 years.
* Patients with the minimum of 5 years of education.
* Patients within the age range of 18 to 35 years.
* Competent and willing to give informed consent.
* Patients living in the study catchment area.

Exclusion Criteria:

* Patients with drug induced psychosis.
* Patients with severe psychopathology, unable to give informed consent.
* Patients suffering from organic or neurological disorder.
* Patients suffering from chronic physical condition.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
50 participant with schizophrenia assessed by PANSS | 2 hours
  30 item question ask from participant
50 participant with schizophrenia assessed by SAI | 30 mintus
  three question each have two parts
50 participant with schizophrenia assessed by PSRS | 1 hour
  6 item on delusion and 11 item on auditory hallucination

REFERENCES:
- [Background] Aleman A, Agrawal N, Morgan KD, David AS. Insight in psychosis and neuropsychological function: meta-analysis. Br J Psychiatry. 2006 Sep;189:204-12. doi: 10.1192/bjp.189.3.204. PMID 16946354
- [Background] Naeem F, Saeed S, Irfan M, Kiran T, Mehmood N, Gul M, Munshi T, Ahmad S, Kazmi A, Husain N, Farooq S, Ayub M, Kingdon D. Brief culturally adapted CBT for psychosis (CaCBTp): A randomized controlled trial from a low income country. Schizophr Res. 2015 May;164(1-3):143-8. doi: 10.1016/j.schres.2015.02.015. Epub 2015 Mar 8. PMID 25757714